CLINICAL TRIAL: NCT06690645
Title: The Association of Psychological Stress with the Efficacy of Neoadjuvant Therapy in Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Director of oncology, Shengjing Hospital
Other Study IDs: MUKDEN-STRESS
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: psychological stress, breast cancer
MeSH Terms: conditions — Breast Neoplasms; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood, tumor tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Exposure: psychological stress status — The assessment of depressive, anxiety or perceived Stress was conducted using PHQ-9, GAD-7 or PSS scale. Patients with a PHQ-9 score ≥ 5 or a GAD-7 score ≥ 5 or a PSS score ≥ 20 were categorized as the stressed group.

SUMMARY:
This study aims to explore the relationship between psychological stress and the therapeutic response in breast cancer patients who have received standard neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumor among women. Approximately 19% to 30% of patients with breast cancer achieve a pathological complete response (pCR) following neoadjuvant therapy, while about 5% to 20% of patients experience disease progression. Increasing evidence suggests the significant role of psychological factors in influencing cancer treatment outcomes. Cancer patients often experience emotional distress, including fear of relapse, anxiety, depression, and low self-esteem, which may persist for many years. Statistics indicate that the incidence of anxiety and depression among cancer patients is 49.69% and 54.90%, respectively, significantly higher than that of healthy individuals (anxiety: 18.37%, depression: 17.50%) in China. There are indications that emotional issues may be linked to cancer treatment, although the underlying mechanisms remain unclear.

This study aims to investigate the relationship between anxiety and depression and the effectiveness of standard neoadjuvant therapy in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥ 18 years; 2.Histological and/or cytological diagnosis of breast cancer; 3.Treatment niave patients; 4.To receive standard neoadjuvant therapy; 5.Eastern Cooperative Oncology Group (ECOG) performance status of 0-1; 6.Presence of at least one measurable lesion according to the Response Evaluation Criteria in Advanced Solid Tumors version 1.1 (RECIST v1.1) ; 7.Informed and agreed to participate in the study;

Exclusion Criteria:

* 1. Breast cancer has not been confirmed through histological or cytological examinations.

  2.Other breast cancer conditions that do not receive neoadjuvant therapy. 3.Combined with other malignant tumors. 4.Concurrent acute or chronic psychiatric disorders, along with having received antidepressant or anti-anxiety therapy within the past month.

  5.Participants must not have engaged in any other clinical trials in the past month, unless those trials are observational or non-interventional in nature.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants included patients diagnosed with breast cancer who were about to receive neoadjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate | 2 years
  pCR is defined as the absence of viable tumor cells in both the tumor bed and lymph nodes. The pCR rate refers to the percentage of patients who achieve this complete response.

SECONDARY OUTCOMES:
Quality of life | 2 years
  Quality of Life (QoL) is assessed using the Functional Assessment of Cancer Therapy-Breast (FACT-B, Version 4.0).
peripheral stress biomarkers | 2 years
  The stress biomarkers, including cortisol and adrenocorticotropic hormone (ACTH), were measured to evaluate the association between peripheral stress biomarkers and the efficacy of neoadjuvant therapy.
Objective Response Rate (ORR) | 2 years
  The objective response rate refers to the proportion of patients whose tumor volume has decreased to a predetermined value and who can maintain that reduction for the minimum required duration.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No